CLINICAL TRIAL: NCT05450237
Title: Psychometric Evaluation in Patients With Brain Damage During Neuroinflammation
Status: Enrolling by invitation | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Diego Centonze, Full Professor, Neuromed IRCCS
Other Study IDs: Punto 5 O.d.g. 30.06.2022
Record Dates: First submitted 2022-07-01; First posted 2022-07-08 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis; Epilepsy; Parkinson Disease; Dementia; Stroke
MeSH Terms: conditions — Multiple Sclerosis; Epilepsy; Parkinson Disease; Dementia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Psychometric Evaluations — The main evaluation scales we will use are the Beck Depression Inventory-II (BDI II), the State-Trait Anxiety Inventory (STAI), The twenty-item Toronto Alexithymia scale- I (TAS-20), The fatigue severity scale (FSS), Modified Fatigue Impact Scale (MFIS), The Multiple Sclerosis Impact Scale (MSIS-29), The Epworth Sleepiness Scale (ESS) (Johns MW. 1991), The Pittsburgh Sleep Quality Index (PSQ1), The Multiple Sclerosis quality of life Inventory (MSQOLI), The work productivity and activity impairment instrument (WPAI), Frailty Index.
  These rating scales will be administered in person, by telephone and / or by sending them electronically.

SUMMARY:
The presence of a damage to the central and / or peripheral nervous system resulting from diseases of a different nature (such as, Multiple Sclerosis, Parkinson's disease, dementia, head trauma, stroke, epilepsy or other neurological syndromes) is commonly cause of both physical than mental disability. The evaluation of certain domains may be more difficult so, specific assessment tools are necessary to analyze them.

DETAILED DESCRIPTION:
The presence of a damage to the central and / or peripheral nervous system resulting from diseases of a different nature (such as, Multiple Sclerosis, Parkinson's disease, dementia, head trauma, stroke, epilepsy or other neurological syndromes) is commonly cause of both physical than mental disability. The presence of cognitive deficits in the sphere of memory or language is often evident at a first clinical examination. However, the evaluation of certain domains such as mood disorders, behavior, sleep-wake cycle or eating habits, may be less evident, even if they have a very strong impact on the quality of life of patients. Specific assessment tools are therefore needed such as psychometric tests, to collect information and analyze the results.

The main evaluation scales we will use are the Beck Depression Inventory-II (BDI II), the State-Trait Anxiety Inventory (STAI), The twenty-item Toronto Alexithymia scale- I (TAS-20), The fatigue severity scale (FSS), Modified Fatigue Impact Scale (MFIS), The Multiple Sclerosis Impact Scale (MSIS-29), The Epworth Sleepiness Scale (ESS), The Pittsburgh Sleep Quality Index (PSQ1), The Multiple Sclerosis quality of life Inventory (MSQOLI), The work productivity and activity impairment instrument (WPAI), Frailty Index.

These rating scales will be administered in person, by telephone and / or by sending them electronically.

ELIGIBILITY:
Inclusion Criteria:

* Presence of brain damage resulting from: Multiple Sclerosis, Parkinson's Disease, Dementia, head trauma, neurosurgery, Stroke, Epilepsy or other neurological syndromes (for the experimental group only);
* Be able to perform the tests to be administered for the duration of the study;
* Patients must be able to follow protocol directions throughout the study;
* Patients must be able to understand the purpose of the study;
* Signature of informed consent, approved by our Ethics Committee.

Exclusion Criteria:

* Inability, even partial, to understand and want;
* Patients with other pathologies that in the opinion of the scientific responsible prevent their recruitment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in follow-up at IRCSS Neuromed in Pozzilli (IS).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
500 patients will be enrolled in the study. The aim is to monitor over time items such as lifestyle indicators, cognitive, functional, emotional abilities and anxiety in patients with various types of neurological damage through use of evaluation scales. | These scales will be administered after certain time intervals. The results obtained will be compared in other to highlight a variation in the scores in the various items.The duration of administration of the scales is approximately one hour.
  The main scales used are:
  * BDI II: evaluates depression during the last week;
  * STAI 1-2: evaluate state anxiety and trait anxiety.
  * TAS-20 is a 20-item questionnaire used to assess alexithymia.
  * FSS: evaluetes the severity of symptoms related to fatigue
  * MFIS: lists 21 items describing the effects of fatigue in relation to their frequency over a four-week period.
  * MSIS-29:evaluates the impact of multiple sclerosis on daily life taking into consideration a time interval of 14 days.
  * ESS: evaluates the likelihood of daytime sleepiness in certain situations, regardless of fatigue.
  * PSQI:investigates the quality of sleep over the past month.
  * MSQOL / 54: evaluates the impact of the disease on the quality of life.
  * WPAI: is a tool that measures the difficulties in work and daily activities due to illness.

CONTACTS AND LOCATIONS:
Overall Officials: Centonze, Principal Investigator — IRCSS Neuromed
Locations (1):
- Ircss Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Hobart J, Lamping D, Fitzpatrick R, Riazi A, Thompson A. The Multiple Sclerosis Impact Scale (MSIS-29): a new patient-based outcome measure. Brain. 2001 May;124(Pt 5):962-73. doi: 10.1093/brain/124.5.962. PMID 11335698
- [Result] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Result] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Result] Larson RD. Psychometric properties of the modified fatigue impact scale. Int J MS Care. 2013 Spring;15(1):15-20. doi: 10.7224/1537-2073.2012-019. PMID 24453758
- [Result] Mitnitski AB, Mogilner AJ, Rockwood K. Accumulation of deficits as a proxy measure of aging. ScientificWorldJournal. 2001 Aug 8;1:323-36. doi: 10.1100/tsw.2001.58. PMID 12806071
- [Result] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Result] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530